CLINICAL TRIAL: NCT05512130
Title: Sodium-Glucose Cotransporter-2 Inhibitors: A Potential Novel Treatment for Epilepsy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FBJH Grant ID 5936
Record Dates: First submitted 2022-07-05; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded, crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin / Placebo (Experimental): Participants randomized to this arm will receive 25 mg of empagliflozin daily for 2 weeks followed placebo daily for 2 weeks
  Interventions: Drug: Empagliflozin 25 mg; Drug: Placebo
- Placebo / Empagliflozin (Experimental): Participants randomized to this arm will receive placebo daily for 2 weeks followed by 25 mg of empagliflozin daily for 2 weeks
  Interventions: Drug: Empagliflozin 25 mg; Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 mg — Participants will take empagliflozin daily for 2 weeks.
  Other Names: Jardiance
Drug: Placebo — Participants will take a placebo daily for 2 weeks. The placebo will be identical to empagliflozin in appearance.

SUMMARY:
About 30% of persons with epilepsy have seizures that do not respond to drugs. The ketogenic diet is an effective treatment option for them, but this high fat diet is strict and difficult to maintain. The properties of gliflozins, which often are used to treat type 2 diabetes, make them a potential replacement for the ketogenic diet. This pilot study will determine whether gliflozins induce ketosis and could be used to treat adults with epilepsy safely.

DETAILED DESCRIPTION:
The 30% of persons with epilepsy who are drug-resistant bear most of the financial and psychosocial costs of this common neurological disorder. An effective, clinically used treatment for these individuals is the ketogenic diet, a high fat, low carbohydrate diet. Newer variants of the ketogenic diet including the modified Atkins diet (MAD) and low glycemic index treatment (LGIT) are more palatable than the older versions but are challenging to maintain because they are strict. The MAD and LGIT lower blood glucose and produce mild ketosis. Sodium-glucose cotransporter-2 inhibitors (SGLT2i) such as empagliflozin have become important additions to the armamentarium for treating type 2 diabetes. SGLT2i decrease blood sugar by causing glucosuria, and they induce mild ketosis. These actions raise the possibility that SGLT2i can replace the MAD and LGIT as epilepsy treatments. This pilot, phase 1 study will determine the feasibility, safety, and tolerability of the SGLT2i empagliflozin in adults with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Focal, generalized, combined generalized and focal, or unknown epilepsy type
* Drug-responsive or drug-resistant epilepsy

Exclusion Criteria:

* Seizure frequency >2 seizures per day during the 6 months prior to enrollment
* Status epilepticus during the 2 years prior to enrollment
* Taking a gliflozin
* Allergy to gliflozins
* Taking a carbonic anhydrase inhibitor such as acetazolamide
* On any ketogenic diet variant
* Having an absolute contraindication to a ketogenic diet
* Type 1 or type 2 diabetes
* Pregnancy
* Moderate to severe intellectual disability,
* Significant cardiovascular disease
* Renal insufficiency
* Body mass index <18.5 or ≥30
* Hemoglobin A1c ≥5.7%

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood beta-hydroxybutyrate while on empagliflozin | 2 weeks
  For each participant, calculate the difference between the blood beta-hydroxybutyrate after two weeks on empagliflozin and after two weeks on placebo.
Change in blood glucose while on empagliflozin | 2 weeks
  For each participant, calculate the difference between the blood glucose after two weeks on empagliflozin and after two weeks on placebo.
Number of participants with adverse effects from empagliflozin | 2 weeks
  For each participant, calculate the difference in weight, blood pressure, and pulse after two weeks on empagliflozin and after two weeks on placebo. Compare the number of participants having an abnormal complete blood count, comprehensive metabolic panel, hemoglobin A1c, magnesium, phosphorus, and urinalysis after two weeks on empagliflozin and after two weeks on placebo. Compare the number of participants who have increased urination and genital irritation after two weeks on empagliflozin and after two weeks on placebo. Will determine the number of participants with a clinically significant change in any of the listed parameters after two weeks on empagliflozin.

SECONDARY OUTCOMES:
Change in seizure frequency | 2 weeks
  For each participant, calculate the difference in seizure frequency as determined by seizure diaries during the two weeks on empagliflozin and the two weeks on placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Kwee L Thio, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all de-identified data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For 3 years beginning one year after study closure
Access Criteria: Qualified investigators upon request.

REFERENCES:
- [Background] Kossoff EH, Krauss GL, McGrogan JR, Freeman JM. Efficacy of the Atkins diet as therapy for intractable epilepsy. Neurology. 2003 Dec 23;61(12):1789-91. doi: 10.1212/01.wnl.0000098889.35155.72. PMID 14694049
- [Background] Pfeifer HH, Thiele EA. Low-glycemic-index treatment: a liberalized ketogenic diet for treatment of intractable epilepsy. Neurology. 2005 Dec 13;65(11):1810-2. doi: 10.1212/01.wnl.0000187071.24292.9e. PMID 16344529
- [Background] Rho JM, Sankar R. The ketogenic diet in a pill: is this possible? Epilepsia. 2008 Nov;49 Suppl 8(Suppl 8):127-33. doi: 10.1111/j.1528-1167.2008.01857.x. PMID 19049610
- [Background] Stafstrom CE, Roopra A, Sutula TP. Seizure suppression via glycolysis inhibition with 2-deoxy-D-glucose (2DG). Epilepsia. 2008 Nov;49 Suppl 8:97-100. doi: 10.1111/j.1528-1167.2008.01848.x. PMID 19049601
- [Background] Stafstrom CE, Ockuly JC, Murphree L, Valley MT, Roopra A, Sutula TP. Anticonvulsant and antiepileptic actions of 2-deoxy-D-glucose in epilepsy models. Ann Neurol. 2009 Apr;65(4):435-47. doi: 10.1002/ana.21603. PMID 19399874
- [Background] Ferrannini E, Baldi S, Frascerra S, Astiarraga B, Heise T, Bizzotto R, Mari A, Pieber TR, Muscelli E. Shift to Fatty Substrate Utilization in Response to Sodium-Glucose Cotransporter 2 Inhibition in Subjects Without Diabetes and Patients With Type 2 Diabetes. Diabetes. 2016 May;65(5):1190-5. doi: 10.2337/db15-1356. Epub 2016 Feb 9. PMID 26861783
- [Background] Kossoff EH, Zupec-Kania BA, Auvin S, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Cross JH, Dahlin MG, Donner EJ, Guzel O, Jehle RS, Klepper J, Kang HC, Lambrechts DA, Liu YMC, Nathan JK, Nordli DR Jr, Pfeifer HH, Rho JM, Scheffer IE, Sharma S, Stafstrom CE, Thiele EA, Turner Z, Vaccarezza MM, van der Louw EJTM, Veggiotti P, Wheless JW, Wirrell EC; Charlie Foundation; Matthew's Friends; Practice Committee of the Child Neurology Society. Optimal clinical management of children receiving dietary therapies for epilepsy: Updated recommendations of the International Ketogenic Diet Study Group. Epilepsia Open. 2018 May 21;3(2):175-192. doi: 10.1002/epi4.12225. eCollection 2018 Jun. PMID 29881797
- [Background] Biester T, Kordonouri O, Danne T. Beyond type 2 diabetes: sodium glucose co-transporter-inhibition in type 1 diabetes. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:53-61. doi: 10.1111/dom.13659. PMID 31081591
- [Background] Kim SR, Lee SG, Kim SH, Kim JH, Choi E, Cho W, Rim JH, Hwang I, Lee CJ, Lee M, Oh CM, Jeon JY, Gee HY, Kim JH, Lee BW, Kang ES, Cha BS, Lee MS, Yu JW, Cho JW, Kim JS, Lee YH. SGLT2 inhibition modulates NLRP3 inflammasome activity via ketones and insulin in diabetes with cardiovascular disease. Nat Commun. 2020 May 1;11(1):2127. doi: 10.1038/s41467-020-15983-6. PMID 32358544